CLINICAL TRIAL: NCT03204279
Title: A Multicenter Multinational Randomized Double Blind PK/PD Dose-finding Study of Oral Netupitant Given With Oral Palonosetron in Pediatric Cancer Patients for Prevention of Nausea and Vomiting Associated With Emetogenic Chemotherapy
Brief Title: PK/PD Study of Netupitant and Palonosetron in Pediatric Patients for Prevention of Chemotherapy-induced Nausea and Vomiting
Acronym: CINV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NEPA-15-31
Record Dates: First submitted 2017-06-14; First posted 2017-07-02 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2020-12

CONDITIONS: Chemotherapy-induced Nausea and Vomiting (CINV)
MeSH Terms: conditions — Vomiting | interventions — netupitant; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Netupitant 1.33 mg/kg plus Palonosetron (Experimental): Single oral dose of Netupitant 1.33 mg/kg up to a maximum of 100 mg (for patients < 3 months of age the netupitant dose will be 0.8 mg/kg) administered with single oral dose of 20 μg/kg palonosetron up to a maximum of 1.5 mg.
  Interventions: Drug: Netupitant; Drug: Palonosetron
- Netupitant 4 mg/kg plus Palonosetron (Experimental): Single oral dose of Netupitant 4 mg/kg up to a maximum of 300 mg (for patients < 3 months of age the netupitant dose will be 2.4 mg/kg) administered with single oral dose 20 μg/kg palonosetron up to a maximum of 1.5 mg.
  Interventions: Drug: Netupitant; Drug: Palonosetron

INTERVENTIONS:
Drug: Netupitant — Netupitant 1.33 mg/kg oral suspension up to a maximum of 100 mg
  Arms: Netupitant 1.33 mg/kg plus Palonosetron
Drug: Palonosetron — Palonosetron 20 μg/kg solution for oral use up to a maximum of 1.5 mg
  Arms: Netupitant 1.33 mg/kg plus Palonosetron
Drug: Netupitant — Netupitant 4 mg/kg oral suspension up to a maximum of 300 mg
  Arms: Netupitant 4 mg/kg plus Palonosetron
Drug: Palonosetron — Palonosetron 20 μg/kg solution for oral use up to a maximum of 1.5 mg
  Arms: Netupitant 4 mg/kg plus Palonosetron

SUMMARY:
This study is Phase 2 pharmacokinetic (PK) and pharmacodynamic (PD) dose-finding study of oral netupitant administered concomitantly with oral palonosetron in pediatric cancer patients for the prevention of nausea and vomiting associated with emetogenic chemotherapy. Two different netupitant dosages will be tested in patients aged from 3 months to < 18 years: 1.33 mg/kg up to a maximum of 100 mg, and 4 mg/kg up to a maximum of 300 mg. All netupitant doses in all age classes will be concomitantly administered with palonosetron 20 μg/kg (up to a maximum dose of 1.5 mg) which is the IV palonosetron dose approved by USA FDA for the pediatric population. The primary objective is to investigate the PK/PD relationship between netupitant exposure (AUC, Cmax) and antiemetic efficacy (CR in delayed phase) after a single oral netupitant administration, concomitantly with oral palonosetron in pediatric cancer patients receiving Moderately Emetogenic Chemotherapy (MEC) or Highly Emetogenic Chemotherapy (HEC) cycles. Efficacy parameter to be used in the correlation is the proportion of patients with Complete Response (CR i.e., no emetic episodes and no rescue medication) during (> 24-120 h after the start of chemotherapy on Day 1).

The secondary objectives are to assess the safety and tolerability after single oral administration of netupitant given concomitantly with a single oral administration of palonosetron; to evaluate the pharmacokinetic (AUC, Cmax, tmax and t1/2) of oral palonosetron at the fixed dose of 20 μg/kg in pediatric patients with the concomitant administration of netupitant. A total of 92 pediatric cancer patients receiving either HEC or MEC will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent by parent(s)/legal guardians of the pediatric patient in compliance with the local laws and regulations. In addition signed children's assent form according to local requirements.
2. Male or female in- or out-patient from birth to < 18 years at the time of randomization.
3. Patient weight at least 3.3 kg.
4. Naïve or non-naïve patient with histologically, and/or cytologically (or imaging in the case of brain tumors) confirmed malignant disease.
5. Scheduled and eligible to receive at least one moderately or highly emetogenic chemotherapeutic agent on Day 1 only or for multiple days.
6. For patient aged ≥ 10 years: Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2.
7. For patient aged 2 years with known mild to moderate hepatic impairment: in the Investigator's opinion the impairment does not jeopardize patient's safety during the study.
8. For patient aged 2 years with known mild to moderate renal impairment: in the Investigator's opinion the impairment should not jeopardize patient's safety during the study.
9. For patient with known history or predisposition to cardiac abnormalities: in the Investigator's opinion the history/predisposition should not jeopardize patient's safety during the study.
10. If the patient is female, she shall: a) not have attained menarche yet or b) have attained menarche and have a negative pregnancy test at the screening visit and at Day 1.
11. Male or female fertile patient using reliable contraceptive measures (such measures, for patient and sexual partner, include: implants, injectables, combined oral contraceptives, intrauterine devices, vasectomized/sterilized partner, use of a double-barrier method or sexual abstinence). The patient and his/her parent(s)/legal guardians must be counseled on the importance of avoiding pregnancy before or during the study.

Exclusion Criteria:

1. The patient and/or parents/caregivers are expected by the Investigator to be non-compliant with the study procedures.
2. Patient has received or is scheduled to receive total body irradiation, total nodal irradiation, upper abdomen radiotherapy, half or upper body irradiation, radiotherapy of the cranium, craniospinal regions, head and neck, lower thorax region or the pelvis within 1 week prior to study entry (Day 1) or within 120 h after start of chemotherapy administration on Day 1.
3. Known history of allergy to any component or other contraindications to any Neurokinin-1 (NK1) or 5-hydroxytryptamine 3 (5-HT3) receptor antagonists.
4. Active infection.
5. Uncontrolled medical condition (e.g., uncontrolled insulin dependent diabetes mellitus).
6. Patient suffering from ongoing vomiting from any organic etiology (including patients with history of gastric outlet obstruction or intestinal obstruction due to adhesions or volvulus, patients with a symptomatic central nervous system(CNS) tumor causing nausea and/or vomiting) or patient with hydrocephalus.
7. Patient who experienced any vomiting, retching, or nausea within 24 h prior to the administration of the study drug
8. Patient who received any drug with potential anti-emetic effect within 24 h prior to the start of reference chemotherapy, including but not limited to:

   NK1- receptor antagonists (e.g., aprepitant or any other new drug of this class); 5-HT3 receptor antagonists (e.g., ondansetron, granisetron, dolasetron, tropisetron, ramosetron); Benzamides (e.g., metoclopramide, alizapride); Phenothiazines (e.g., prochlorperazine, promethazine, perphenazine, fluphenazine, chlorpromazine, thiethylperazine); Benzodiazepines initiated 48 h prior to study drug administration or expected to be received within 120 h following initiation of chemotherapy, except for single doses of midazolam, temazepam or triazolam; Butyrophenones (e.g., droperidol, haloperidol); Anticholinergics (e.g., scopolamine, with the exception of inhaled anticholinergics for respiratory disorders e.g., ipratropium bromide); Antihistamines (e.g., diphenhydramine, cyclizine, hydroxyzine, chlorpheniramine, dimenhydrinate, meclizine); Domperidone; Mirtazapine; Olanzapine; Prescribed cannabinoids (e.g., tetrahydrocannabinol, nabilone); Over the Counter (OTC) antiemetics, OTC cold or OTC allergy medications; Herbal preparations containing ephedra or ginger.
9. Patient who received palonosetron within 1 week prior to administration of study drug.
10. Patient who has been started on systemic corticosteroid therapy within 72 h prior to study drug administration or is planned to receive a corticosteroid as part of the chemotherapy regimen
11. Patient aged < 6 years who received any investigational drug (defined as a medication with no marketing authorization granted for any age class and any indication) within 90 days prior to Day 1, or patient aged 6 years who received any investigational drug within 30 days prior to Day 1 or is expected to receive investigational drugs prior to study completion.
12. Intake of alcohol, food or beverages (e.g., grapefruit, cranberry, pomegranate and aloe vera juices, German chamomile) known to interfere with either CYP3A4 or CYP2D6 metabolic enzymes within 1 week prior to Day 1 and during the overall study period.
13. Use of any drugs or substances known to be strong or moderate inhibitors of CYP3A4 and CYP2D6 enzymes within 1 week prior to Day 1 or planned to be used during the overall study period.
14. Use of any drugs or substances known to be CYP3A4 substrates with narrow therapeutic range within 1 week prior to Day 1, or planned to be used during the overall study period.
15. Use of any drugs or substances known to be inducers of CYP3A4 enzymes within 4 weeks prior to Day 1 or planned to be used during the overall study period.
16. Lactating female patient.
17. Patient with clinically relevant abnormal laboratory values that in the Investigator's opinion jeopardize the patient's safety during the study.
18. Patient aged < 2 years with known hepatic impairment (any grade), or patient aged 2 years with known severe hepatic impairment.
19. Patient aged < 2 years with known renal impairment (any grade), or patient aged 2 years with known severe renal impairment.
20. Enrolment in a previous study with netupitant (either alone or in combination with palonosetron).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - Nemours/A.I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Hospital - Orlando, Orlando, Florida
  - Maine Medical Center - Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Medical University of South Carolina, Charleston, South Carolina
- Russia (7):
  - Chelyabinsk Regional Children's Clinical Hospital, Chelyabinsk
  - Children's Territorial Clinical Hospital, Krasnodar
  - Dmitry Rogachev National Scientific and Practical Center for Pediatric Hematology, Oncology and Immunology, Moscow
  - City Clinical Hospital #31, Saint Petersburg
  - First I.P. Pavlov State Medical University of St. Petersburg, Saint Petersburg
  - Voronezh Regional Children's Cinical Hospital #1, Voronezh
  - Regional Children's Clinical Hospital #1, Yekaterinburg
- Serbia (2):
  - University Children's Hospital, Center for Pediatrics, Department of Hematology and Oncology, Belgrade
  - Clinical Center Nis, Clinic of Pediatric Internal Diseases, Niš
- Ukraine (3):
  - Dnipropetrovsk Regional Children's Clinical Hospital, Dnipro
  - National Institute of Cancer, Research Department of Pediatric Oncology, Kyiv
  - West Ukrainian Specialized Children's Medical Center, Department of Pediatric Surgery, Lviv

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron | Netupitant 4 mg/kg Plus Palonosetron
Started | 34 | 33
Completed | 34 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Male and female pediatric cancer patients from birth up to <18 years, who were scheduled to receive HEC or MEC to be administered as single-day chemotherapy on Day 1 only or for multiple days. All participants who received study drug. In netupitant 4 mg/kg arm 1 patient was withdrew from the study after randomization of study drug and was not treated with the study drug (the overall number of participants started in netupitant 4 mg/kg arm was 33 and 32 patients completed the study).
Groups:
- Total: Total of all reporting groups
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron | Netupitant 4 mg/kg Plus Palonosetron | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (6.29) | 5.6 (5.46) | 6.1 (5.88)
Age, Customized [Count of Participants; unit: Participants]
  3 to <6 months | 3 | 2 | 5
  6 to <12 months | 4 | 5 | 9
  1 to <2 years | 3 | 4 | 7
  2 to <5 years | 6 | 6 | 12
  5 to <12 years | 8 | 8 | 16
  12 to <18 years | 9 | 7 | 16
  1 to <3 months | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 21 | 18 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 31 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of Netupitant
Description: Mean values of area under the plasma Concentration versus time curve from time zero to infinity (AUC0-inf) of netupitant after a single oral netupitant administration, concomitantly with oral palonosetron, in pediatric cancer patients receiving HEC or MEC cycles. AUC estimates are obtained by non-compartmental analysis of population model-predicted individual plasma concentration-time profiles.
Time Frame: within 168 hours after netupitant administration. A sampling windows approach will be used by collecting a single blood sample from each patient in one of these time windows: from 2 to 8 h, from 24 to 48 h, from 72 to 96 h and from 120 to 168 h.
Population: Pediatric patients divided in seven age groups; in netupitant 4 mg/kg arm 1 patient was withdrew from the study after randomization of study drug and was not treated; 1 patient was treated with study drug but did not receive the entire planned dose and was not included in this analysis and one patient received the entire planned dose, but did not have any measurable concentration of netupitant and/or palonosetron.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron | Netupitant 4 mg/kg Plus Palonosetron
Number analyzed (Participants) | 34 | 30
ng*hr/mL
  patients 1 month to <3 months of age: number analyzed (Participants) | 1 | 0
  patients 1 month to <3 months of age | 4460 |
  patients 3 month to <6 months of age: number analyzed (Participants) | 3 | 2
  patients 3 month to <6 months of age | 3849 (91.3) | 17340 (36.4)
  patients 6 month to <1 year of age: number analyzed (Participants) | 4 | 4
  patients 6 month to <1 year of age | 7637 (113) | 8617 (45.2)
  patients 1 year to <2 years: number analyzed (Participants) | 3 | 4
  patients 1 year to <2 years | 2276 (29.8) | 9886 (59.6)
  patients 2 years to <5 years: number analyzed (Participants) | 6 | 6
  patients 2 years to <5 years | 3135 (44.0) | 14404 (131)
  patients 5 years to <12 years: number analyzed (Participants) | 8 | 8
  patients 5 years to <12 years | 2676 (35.0) | 10154 (70.7)
  patients 12 years to <18 years: number analyzed (Participants) | 9 | 6
  patients 12 years to <18 years | 3107 (54.9) | 12266 (26.9)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Netupitant
Description: Mean values of maximum plasma concentration (Cmax) of netupitant after a single oral netupitant administration, concomitantly with oral palonosetron, in pediatric cancer patients receiving HEC or MEC cycles. Cmax estimates are obtained by non-compartmental analysis of population model-predicted individual plasma concentration-time profiles
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron | Netupitant 4 mg/kg Plus Palonosetron
Number analyzed (Participants) | 34 | 30
ng/mL
  1 month to <3 months: number analyzed (Participants) | 1 | 0
  1 month to <3 months | 60.8 (NA) — For only one measurement CV is not available |
  3 months to <6 months: number analyzed (Participants) | 3 | 2
  3 months to <6 months | 76.0 (27.1) | 233 (4.25)
  6 months to <12 months: number analyzed (Participants) | 4 | 4
  6 months to <12 months | 133 (71.7) | 255 (31.2)
  1 year to <2 years: number analyzed (Participants) | 3 | 4
  1 year to <2 years | 69.5 (19.3) | 275 (38.2)
  2 years to <5 years: number analyzed (Participants) | 6 | 6
  2 years to <5 years | 74.0 (32.3) | 266 (55.0)
  5 years to <12 years: number analyzed (Participants) | 8 | 8
  5 years to <12 years | 67.9 (32.1) | 213 (20.1)
  12 years to <18 years: number analyzed (Participants) | 9 | 6
  12 years to <18 years | 76.8 (27.3) | 274 (15.6)

3. Primary Outcome: Exposure - Response Analysis for Netupitant
Description: Exposure - Response analysis for netupitant performed by assessing the relationships between exposure parameters AUC0-inf and Cmax with the primary efficacy endpoint, i.e., the CR in the delayed phase.
  Graphical exposure-response analysis for netupitant performed by assessing the relationship between individual exposure parameters (AUC0-inf) and Cmax) with the primary efficacy endpoint, i.e the CR in the delayed phase.
Time Frame: > 24-120 hours after the start of chemotherapy on Day 1
Population: All pediatric patients with exposures parameters and CR data in the delayed phase
Measure: Count of Participants; unit: Participants
Groups:
- Netupitant 1.33 mg/kg Plus Palonosetron or Netupitant 4 mg/kg Plus Palonosetron: Single oral dose of Netupitant 1.33 mg/kg up to a maximum of 100 mg (for patients < 3 months of age the netupitant dose will be 0.8 mg/kg) administered with single oral dose of 20 μg/kg palonosetron up to a maximum of 1.5 mg.
  Or Single oral dose of Netupitant 4 mg/kg up to a maximum of 300 mg (for patients < 3 months of age the netupitant dose will be 2.4 mg/kg) administered with single oral dose 20 μg/kg palonosetron up to a maximum of 1.5 mg.
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron or Netupitant 4 mg/kg Plus Palonosetron
Number analyzed (Participants) | 64
Participants
  number of participants with CR in delayed phase | 45
  number of participants with no CR in delayed phase | 19
Statistical Analysis 1: Comparison: Netupitant 1.33 mg/kg Plus Palonosetron or Netupitant 4 mg/kg Plus Palonosetron; The population consist of all patients having CR in the delayed phase and AUC0-inf and Cmax, there is no comparison between the two dose groups; Test type: Other — No comparison between the two dose groups is performed, thus no statistical test is applied. In the next section the goodness of fit of the loess function correlating exposure and response is reported; p = 0.55, loess (Local regression or polynomial) — CR in the delayed phase vs AUC0-inf; The p-value represents the probability found if the correlation coefficient was zero (null hypothesis); Pearson R = 0.076 — R is the Pearson correlation is a coefficient statistic that measures linear correlation between two variables CR in the delayed phase vs AUC0-inf
Statistical Analysis 2: Comparison: Netupitant 1.33 mg/kg Plus Palonosetron or Netupitant 4 mg/kg Plus Palonosetron; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.75, loess (Local regression or polynomial) — CR in the delayed phase vs Cmax; The p-value represents the probability found if the correlation coefficient was zero (null hypothesis); Pearson R = -0.041 — R is the Pearson correlation is a coefficient statistic that measures linear correlation between two variables CR in the delayed phase vs Cmax

4. Secondary Outcome: Percentage of Pediatric Patients With Complete Response During the Delayed Phase
Description: Percentage of Pediatric Patients with complete response (CR, i.e., no emetic episodes and no rescue medication) during the delayed phase (> 24 to 120 h after the start of chemotherapy on Day 1) after a single oral netupitant administration, concomitantly with oral palonosetron, in pediatric cancer patients receiving HEC or MEC cycles.
Time Frame: > 24-120 hours after the start of chemotherapy on Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron | Netupitant 4 mg/kg Plus Palonosetron
Number analyzed (Participants) | 34 | 31
Participants | 24 | 22

ADVERSE EVENTS:
Time Frame: From the first dose of study drug on Visit 2 (Day 1, inclusively) until Visit 5 (follow up, Day 14 [+3])
Arm/Group | Netupitant 1.33 mg/kg Plus Palonosetron | Netupitant 4 mg/kg Plus Palonosetron
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/34 | 3/32
Other Adverse Events (participants affected / at risk) | 22/34 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netupitant 1.33 mg/kg Plus Palonosetron (N=34) | Netupitant 4 mg/kg Plus Palonosetron (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netupitant 1.33 mg/kg Plus Palonosetron (N=34) | Netupitant 4 mg/kg Plus Palonosetron (N=32)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 7 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 8 (8) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 6 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4)
Complication associated with device (General disorders) | 1 (1) | 1 (2)
Pyrexia (General disorders) | 1 (2) | 5 (5)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03204279/Prot_SAP_001.pdf